CLINICAL TRIAL: NCT03459638
Title: Periodontitis as a Potential Early Risk Indicator for Diabetes Mellitus, Atherosclerotic Cardiovascular Disease, Metabolic Syndrome and Obstructive Sleep Apnea Syndrome
Brief Title: Periodontitis as Signal for an Underlying Disease
Acronym: PACMEL
Status: Completed | Type: Observational
Sponsor: Academic Centre for Dentistry in Amsterdam (Other)
Collaborators: Labonovum B.V. (Unknown); Sunstar Suisse S.A. (Unknown); Netherlands Enterprise Agency (Unknown)
Responsible Party: Principal Investigator, M. X. F. Kosho, Principal Investigator, Academic Centre for Dentistry in Amsterdam
Other Study IDs: PerioSystemicACTA
Record Dates: First submitted 2018-03-02; First posted 2018-03-09 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus; Periodontal Diseases; Cardiovascular Diseases; Obstructive Sleep Apnea Syndrome
Keywords: Screening
MeSH Terms: conditions — Diabetes Mellitus; Periodontal Diseases; Cardiovascular Diseases; Sleep Apnea, Obstructive | interventions — Mass Screening; ETV3 protein, human

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood and oral rinse sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Periodontitis: Screening for DM, ASCVD, MetS and OSAS in patients with periodontitis
  Interventions: Other: Screening for DM, ASCVD, MetS and OSAS
- No periodontitis: 'Screening for DM, ASCVD, MetS and OSAS in patients without periodontitis
  Interventions: Other: Screening for DM, ASCVD, MetS and OSAS

INTERVENTIONS:
Other: Screening for DM, ASCVD, MetS and OSAS — Finger stick analysis, questionnaires and clinical measurements

SUMMARY:
This study investigates the differences between subjects with and without periodontitis in: the prevalence of (pre)diabetes mellitus, the risk of atherosclerotic cardiovascular disease, the prevalence of metabolic syndrome and the risk of obstructive sleep apnea syndrome.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM), Atherosclerotic Cardiovascular Disease (ASCVD), Metabolic Syndrome (MetS) and Obstructive Sleep Apnea Syndrome (OSAS) are major health problems. However due to absence of symptoms and/or lack of knowledge, people are often unaware of having DM, ASCVD, MetS or OSAS while early treatment could prevent or stop the progression of these diseases. Therefore risk indicators for early detection of DM, ASCVD, MetS and OSAS are needed and proposed.

Many studies demonstrate the association between oral diseases and DM and/or ASCVD. The most observed chronic oral disease is periodontitis. Periodontitis is a common chronic multifactorial inflammatory disease of the supporting structures of the teeth. DM and ASCVD might, due to their proinflammatory state and alteration of the immune system, contribute to the onset and/or progression of periodontitis. Therefore periodontitis could be considered as an early sign of an underlying vascular and/or metabolic pathology.

Some studies have also reported a positive association between periodontitis and MetS. The MetS prevalence in patients with periodontitis was shown to be higher than controls and MetS showed to be associated with severe periodontitis. The association between periodontitis and OSAS is less established, however there is some evidence to a plausible association between periodontal disease and Obstructive Sleep Apnea (OSA).

Due to the broad overlap of objective biomarkers, in this study, subjects with or without periodontitis will be screened for determining the prevalence of (pre)DM, the 10 year risk of ASCVD, the prevalence of MetS and the risk of OSAS.

The screening will be based on clinical measures, specific blood markers determined by a developed finger stick procedure and three questionnaires.

Notably, a recently published pilot paper from the ACTA periodontology research group presents the feasibility and preliminary results of proposed screening for (pre)DM; 18.1% new DM cases were found among subjects with severe periodontitis, compared to 9.9% in mild/moderate periodontitis and 8.5% in controls.

Objective of the study:

The aim of the proposed study is to screen for (pre)DM, an increased 10 year risk of ASCVD, MetS and a high risk of OSAS in participants with and without periodontitis. Consequently, the dental office will be evaluated as a suitable location for early detection of these diseases.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, a subject must meet all of the following criteria:
* Age ≥ 40 years
* (Patient) referred for periodontitis
* (Control) visiting the dental school for regular dental check-up without periodontitis
* Able and willing to give written informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: : In total 200 patients will be included at the Academic Centre for Dentistry Amsterdam (ACTA). The subjects with periodontitis that will be enrolled in this study are referred to the periodontal clinic for diagnosis and treatment of periodontitis. The subjects without periodontitis will be selected among individuals that visit the dental school for regular dental checkups. All subjects will be 40 years and older and are mainly inhabitants from Amsterdam and surrounding areas.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of prediabetes and diabetes (DM) | 24 months
  For DM there is the convenient Haemoglobin A1c (HbA1c) level, which is put forward by the American Diabetes Association (ADA) and International Diabetes Federation (IDF) as indicative of the metabolic state: prediabetes (HbA1c: 39-47 mmol/mol) and diabetes (HbA1c: ≥48 mmol/mol).
10-year-risk of atherosclerotic cardiovascular disease (ASCVD) | 24 months
  For ASCVD there is the "10-year-risk" chart, based on age, gender, total cholesterol, HDL cholesterol (HDL-C), LDL cholesterol (LDL-C), systolic and diastolic blood pressure, smoking, presence of diabetes and rheumatoid arthritis (according to the NHG standards, which are the European Society of Cardiology guidelines modified to the Dutch population). The 10-year risk of death or disease by ASCVD can be: Low = <10%, Middle = 10-20%, High = >20%.
Prevalence of metabolic syndrome (MetS) | 24 months
  The diagnostic criteria for MetS are based on the waist circumference (WC), triglycerides (TG), HDL-C, hypertension and dysglycemia (according to the NCEP ATP III). Any 3 of these 5 measures constitute diagnosis of metabolic syndrome. The outcome will be: 1. Absence of MetS (when ≤ 2 measures are met for the criteria of MetS) ; 1. Presence of MetS (when ≥ 3 measures are met for the criteria of MetS).
Risk of obstructive sleep apnea syndrome (OSAS) | 24 months
  For OSAS there is the recently developed OSAS risk questionnaire (Philips questionnaire), which scores patients into a low, high or severe risk category of having OSAS.The outcome will be on a percentage scale, varying from 0-100%. The cut-off point for being classified into the low risk category will be 35% and the cutt-of point for the severe risk category is 55%. Between 35 and 55%, participants are classified as high risk for OSAS.

CONTACTS AND LOCATIONS:
Overall Officials: Madeline X. F. Kosho, MSc, DDS, Principal Investigator — Academic Centre for Dentistry Amsterdam
Locations (1):
- Academic Centre for Dentistry Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Teeuw WJ, Kosho MX, Poland DC, Gerdes VE, Loos BG. Periodontitis as a possible early sign of diabetes mellitus. BMJ Open Diabetes Res Care. 2017 Jan 19;5(1):e000326. doi: 10.1136/bmjdrc-2016-000326. eCollection 2017. PMID 28316794
- [Background] Nibali L, Tatarakis N, Needleman I, Tu YK, D'Aiuto F, Rizzo M, Donos N. Clinical review: Association between metabolic syndrome and periodontitis: a systematic review and meta-analysis. J Clin Endocrinol Metab. 2013 Mar;98(3):913-20. doi: 10.1210/jc.2012-3552. Epub 2013 Feb 5. PMID 23386648
- [Background] Al-Jewair TS, Al-Jasser R, Almas K. Periodontitis and obstructive sleep apnea's bidirectional relationship: a systematic review and meta-analysis. Sleep Breath. 2015 Dec;19(4):1111-20. doi: 10.1007/s11325-015-1160-8. Epub 2015 Mar 24. PMID 25801281
- [Background] Friedewald VE, Kornman KS, Beck JD, Genco R, Goldfine A, Libby P, Offenbacher S, Ridker PM, Van Dyke TE, Roberts WC; American Journal of Cardiology; Journal of Periodontology. The American Journal of Cardiology and Journal of Periodontology editors' consensus: periodontitis and atherosclerotic cardiovascular disease. J Periodontol. 2009 Jul;80(7):1021-32. doi: 10.1902/jop.2009.097001. PMID 19563277
- [Background] Beukers NG, van der Heijden GJ, van Wijk AJ, Loos BG. Periodontitis is an independent risk indicator for atherosclerotic cardiovascular diseases among 60 174 participants in a large dental school in the Netherlands. J Epidemiol Community Health. 2017 Jan;71(1):37-42. doi: 10.1136/jech-2015-206745. Epub 2016 Aug 8. PMID 27502782

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT03459638/Prot_SAP_000.pdf